CLINICAL TRIAL: NCT05634434
Title: Uric Acid Based Renal Stones: Clinical, Metabolic and Genetic Characterization Looking for Determinants of Recurrence and Laterality
Brief Title: Uric Acid Based Renal Stones: Clinical, Metabolic and Genetic Characterization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Assistant Professor of Urology, Mansoura University
Other Study IDs: MS.21.08.1617
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Renal Stone; Urinary Stones
Keywords: kidney stones; uric acid
MeSH Terms: conditions — Nephrolithiasis; Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples were collected from the renal pelvis of the kidney using ureteric catheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Same patient, stone free kidney
- Study group: uric acid stone former, diseased kidney (stone harboring)

SUMMARY:
* Reporting prevalence of uric acid based renal stones among patients with nephrolithiasis admitted to Mansoura Urology and Nephrology center (MUNC).
* Furthermore, identification of monogenic and polygenic uric acid stone formers.
* Identification of factors associated uric acid stone recurrence as well as determinants of laterality in patients with uric acid based renal stones

DETAILED DESCRIPTION:
* To Report the prevalence of uric acid based renal stones among patients with NL admitted to Mansoura Urology and Nephrology center (MUNC).
* To identify monogenic and polygenic uric acid stone formers.
* To Identify the factors associated uric acid stone recurrence as well as determinants of their laterality in patients with uric acid based renal stones.
* Research Approach and Methodology
* Study design: A prospective controlled study
* Target population:

Patients admitted in Mansoura urology and nephrology center with unilateral or bilateral renal stones, as proven by imaging techniques (ultrasound and non-contrast spiral CT scan) are targeted in the duration between September 2021 to September 2022.

Healthy stone free individuals proven by imaging are assigned as a control group.

Legible subjects fulfilling inclusion criteria will be included in a prospective study and will be asked to sign an informed consent form according to Good Clinical Practice and the Declaration of Helsinki.

* Inclusion criteria should satisfy all the following.
* Patients with unilateral or bilateral renal stones (de novo or recurrent) who are candidates for endoscopic treatment (percutaneous nephrolithotomy).
* Patients with preoperative NCCT findings of renal stone with stone density equal or less than 600HU.
* Patients with dominant uric acid composition will be included as proven by postoperative stone analysis.
* Exclusion criteria:
* Patients with anatomical abnormalities precipitating stone disease e.g. ureteric stricture, ureteropelvic or ureterovesical junction obstruction, Urinary diversion, History of ureterovesical re-implantation
* Patients with non-uric acid stones as proven by post-operative stone analysis.
* Study groups
* Control group, Healthy stone free individuals proven by imaging will be assigned as a control group.
* Study group
* Denovo uric acid stone former (DUASF)
* Recurrent uric acid stone former (RUASF)
* Assessment tools
* History includes residence, nutritional history, medical history e.g, DM and its type and history of stone disease +/- previous intervention.
* Exam includes BMI, waist and hip circumference, waist-to-hip ratio, and blood pressure reporting.
* Preoperative work up includes.
* Urine analysis (Dipstick and microscopy)
* 24-hours urine collection for (Ph, ammonium, citrate, urate, and Tamm-Horsfall Protein (THP))
* Blood sample for TLC (neutrophil and lymphocyte count), HgA1c, serum creatinine and uric acid level
* Operative procedure and findings After overnight hydration using physiological saline 0.9% at a rate of 1ml/min. PCNL will be carried out in standard approach with bilateral ureteric catheters insertion.
* Differential urine sampling from each kidney; Separate renal units' drainage with differential urine sampling will be carried out before creation of the renal puncture. Urine will be tested for Ph, ammonium, citrate, urate, and Tamm-Horsfall Protein (THP).
* Stone analysis will be carried out using infrared spectroscopy.
* Genetic testing Genomic DNA will be extracted from peripheral blood leukocytes using standard methods. The primer pairs and PCR reaction conditions that will be designed for used SLC22A12 and SLC2A9 to amplify the sequences. For all PCR reactions, we will use 50 to 100 ng of genomic DNA, 5 to 10 pmol of reverse and forward primers Sequencing will be performed in both directions using the ABI PRISM 3700 DNA Analyzer (Applied Biosystems).
* Postoperative work up, includes before discharge control NCCT to rule out any residual stones. Patients with any non-targeted lucent residuals will be offered oral dissolution therapy in the form of potassium citrate till deemed stone free by NCCT at 3 months. All stone free patients will be advised for general stone preventive measures e.g, plenty of fluid intake and control of serum uric acid level. Patients will be invited for one year follow up visit for NCCT and any recurrent stone will be depicted, and its characters will be assessed in standard way.
* Sample size and data analysis:

All patients with renal stones subjected to PNL will have stone analysis. For genetic, molecular, and metabolic evaluation; control group will be 10 healthy stone free volunteers and study group will include 20 uric acid stone patients.

Data will be collected into IBM SPSS25 program (social package for statistical sciences, IBM Corporation; Armonk, New York, USA). The mean and standard deviation (median and range) of all continuous measures and scores will be reported as indicated. Number (%) for categorical variables if any will be recorded at baseline and all subsequent visits. Proper statistical tests will be utilized accordingly.

* Outcomes:
* The primary outcome: reporting overall prevalence of uric acid stones among patients with renal stones admitted in Mansoura UNC during study period.
* Secondary outcomes, include identification of genetic alterations in patients with uric acid stones and possible correlation with stone recurrence over 1 year following stone clearance. Reporting distinct clinical, metabolic and genetic features among uric acid stone formers with attempt for correlation of these findings to stone laterality.

ELIGIBILITY:
Inclusion Criteria:

* ⦁ Patients with unilateral renal stones (denovo or recurrent) who are candidates for endoscopic treatment (percutaneous nephrolithotomy).

  * Patients with preoperative NCCT findings of renal stone with stone density equal or less than 600HU.
  * Patients with dominant uric acid composition will be included as proven by postoperative stone analysis

Exclusion Criteria:

* ⦁ Patients with anatomical abnormalities precipitating stone disease e.g. ureteric stricture, ureteropelvic or ureterovesical junction obstruction, Urinary diversion, History of ureterovesical re-implantation

  * Patients with non-uric acid stones as proven by post-operative stone analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Uric acid-based renal stone formers
  * Denovo uric acid stone former (DUASF)
  * Recurrent uric acid stone former (RUASF)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
reporting overall prevalence of uric acid stones | 1 year
  reporting overall prevalence of uric acid stones among patients with renal stones admitted in Mansoura UNC during study period.

SECONDARY OUTCOMES:
identification of genetic alterations in patients with uric acid stones | 1year
  identification of genetic alterations in patients with uric acid stones and possible correlation with stone recurrence over 1 year following stone clearance. Reporting distinct clinical, metabolic and genetic features among uric acid stone formers with attempt for correlation of these findings to stone laterality.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided